CLINICAL TRIAL: NCT03880071
Title: Efficacy of a Dialectical Behavior Therapy and Acceptance Commitment Therapy Short Program for Prevention of Suicidal Behavior in Patients With Borderline Personality Disorder
Brief Title: DIalectical Behavior Therapy and Acceptance Commitment Therapy Short Program for BOrderLine persOnality Disorder
Acronym: DIABOLO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Abandoned study
Sponsor: University Hospital, Montpellier (Other)
Collaborators: INSERM 1061, " Neuropsychiatry: epidemiological and clinical research", Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL18_0044
Record Dates: First submitted 2019-03-14; First posted 2019-03-19 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Female; Borderline Personality Disorder
Keywords: Psychiatry; Suicidal Behavior; Borderline Personality Disorder; Prevention; Dialectic Behavioral Therapy; Acceptance Commitment Therapy
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBT + ACT group (Experimental): - The experimental group (DBT+ ACT) led in Montpellier during 6 months.
  Interventions: Behavioral: DBT+ACT
- DBT group (Other): The control group (DBT) led in Geneva during 12 months.
  Interventions: Behavioral: DBT

INTERVENTIONS:
Behavioral: DBT+ACT — - The experimental group (DBT+ ACT) will have: 25 therapy group sessions (1 sessions of 2 hours once a week) 25 individual interview sessions (1 sessions of 1 hour once a week) will receive 25 group sessions and 25 individual ones during 6 months.
  Arms: DBT + ACT group
Behavioral: DBT — The control group (DBT) will have:
  50 therapy group sessions (1 session of 2h30 once a week) 50 individual interview sessions (1 sessions of 1 hour once a week)
  Arms: DBT group

SUMMARY:
According to the World Health Organization 1 death by suicide occurs every 40 seconds, leading suicide prevention to one of the public health priority.

Borderline personality disorder (BPD) is a common condition affecting 6% of the population.

This disorder is characterized by unstable emotions, unstable mood, difficulties with relationship and feer of abandonment.

BPD is also the psychopathology the most related to suicidal attempts. Indeed, up to 50% of the patients admitted to hospital after a suicide attempt are diagnosis with a BPD.

Negative interpersonal events (events occurring between two people) are known as the main stressor that trigger a suicidal attempt.

People with a BPD are highly sensitive to it. Unfortunately, patient care for this disorder is limited. Pharmacological strategies didn't show any efficacy and psychotherapies, although proven effective, are difficult to set up.

As BPD is strongly related to suicidal attempts it appears to be a good model to study suicidal behavior. Thus, this study could improve knowledge in this field.

Suicidal behavior in patients receiving the standard therapy (dialectic behavioural therapy: DBT) will be compared to patients receiving dialectical behavior therapy and acceptance commitment therapy (ACT).

Clinical data reflecting how the participant is feeling will be collected as well.

DETAILED DESCRIPTION:
An emotional dysregulation has been linked to suicidal behavior in patients with BPD.

Up to this date, no program had combined dialectical behavior therapy with acceptance commitment therapy.

DBT aims to teach skills in four different fields : mindfulness, emotional regulation, distress tolerance and interpersonal efficiency.

ACT helps to develop metacognitive skills and to identify what makes sense in one's life.

Because 75% of BPD patients are women, the study will only focus on them.

Patients will be evaluated during 4 visits :

* Inclusion : 1 or 2 weeks before the first session of therapy. During this visit patients will undergo a clinical exam and will complete questionnaires.
* First follow-up visit : 6 months after the first session (for the experimental group) or 12 months after the first session (for the control group). During this visit will undergo a clinical exam and will complete questionnaires. Therapeutic processes, therapy satisfaction and cost- effectiveness ratio will be evaluated
* Second follow-up visit : 12 months after the first sessions (for the experimental group) or 18 months after the first session (for the control group). During this visit will undergo a clinical exam and will complete questionnaires. Therapeutic processes, and cost- effectiveness ratio will be evaluated
* Third follow-up visit : 18 months after the first session (for the experimental group) or 24 months after the first session (for the control group). During this visit will undergo a clinical exam and will complete questionnaires. Therapeutic processes, and cost- effectiveness ratio will be evaluated The hypothesis is that DBT+ ACT allows reducing suicidal recidivism, reducing economical cost linked to BPD and improving quality of life and functioning among patients.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman
* Between 18 and 50 years old
* Clinical diagnosis of BPD using the Structured Clinical Interview for DSM-IV-TR ( Diagnostic and Statistical Manual of mental disorders) Axis II Personality Disorders)
* Having signed the informed consent
* Able to realize all the visits and therapy sessions
* Able to speak, read and understand French

Exclusion Criteria:

* Life time diagnosis of schizophrenia
* Life time diagnosis of intellectual disability
* Not able to read and write
* Refusal of participation
* Subject protected by law (guardianship)
* Deprived of liberty Subject (by judicial or administrative decision)
* Not belonging to social safety system
* Exclusion period in relation to another protocol

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Number of proven suicide attempts using the Columbia-Suicide severity rating scale (C-SSRS) at 1 year follow-up | At 1 year after the intervention
  Evaluation and comparison of suicide attempts number before and after therapy between DBT and DBT+ACT groups with the Columbia-Suicide severity rating scale : indication of the number of proven suicide attempts and score from 0 to 5 depending on the severity of the suicide attempt

SECONDARY OUTCOMES:
Evolution of suicidal symptomatology using the Columbia Suicide Severity Rating Scale (C-SSRS) | At one week after the intervention
  Evaluation and comparison of suicidal symptomatology between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 17 close-ended questions of the Columbia-Suicide severity rating scale
Evolution of suicidal symptomatology using the Columbia Suicide Severity Rating Scale (C-SSRS) | At 6 months after the intervention
  Evaluation and comparison of suicidal symptomatology between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 17 close-ended questions of the Columbia-Suicide severity rating scale
Evolution of suicidal symptomatology using the Columbia Suicide Severity Rating Scale (C-SSRS) | At 12 months after the intervention
  Evaluation and comparison of suicidal symptomatology between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 17 close-ended questions of the Columbia-Suicide severity rating scale
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At one week after the intervention
  Evaluation and comparison of suicidal symptomatology between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At 6 months after the intervention
  Evaluation and comparison of suicidal symptomatology between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At 12 months after the intervention
  Evaluation and comparison of suicidal symptomatology between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal intensity of suicidal intent) | At one week after the intervention
  Evaluation and comparison of intensity of suicidal intent between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal intensity of suicidal intent) | At 6 months after the intervention
  Evaluation and comparison of intensity of suicidal intent between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal intensity of suicidal intent) | At 12 months after the intervention
  Evaluation and comparison of intensity of suicidal intent between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal intensity of imperious need for non-suicidal self-damaging behavior) | At one week after the intervention
  Evaluation and comparison of intensity of imperious need for non-suicidal self-damaging behavior between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal intensity of imperious need for non-suicidal self-damaging behavior) | At 6 months after the intervention
  Evaluation and comparison of intensity of imperious need for non-suicidal self-damaging behavior between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal intensity of imperious need for non-suicidal self-damaging behavior) | At 12 months after the intervention
  Evaluation and comparison of intensity of imperious need for non-suicidal self-damaging behavior between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal quality of perceived social support) | At one week after the intervention
  Evaluation and comparison of quality of perceived social support between pre-intervention and post-intervention (one week after the last session of the intervention)within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal quality of perceived social support) | At 6 months after the intervention
  Evaluation and comparison of quality of perceived social support between pre-intervention and post-intervention (one week after the last session of the intervention)within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal quality of perceived social support) | At 12 months after the intervention
  Evaluation and comparison of quality of perceived social support between pre-intervention and post-intervention (one week after the last session of the intervention)within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal psychological pain) | At one week after the intervention
  Evaluation and comparison of psychological pain between pre-intervention and post-intervention (one week after of the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal psychological pain) | At 6 months after the intervention
  Evaluation and comparison of psychological pain between pre-intervention and post-intervention (one week after of the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal psychological pain) | At 12 months after the intervention
  Evaluation and comparison of psychological pain between pre-intervention and post-intervention (one week after of the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (not all characteristic of my way of being) to 10 (completely characteristic of my way of being) | At one week after the intervention
  Evaluation and comparison of the evolution of intensity of each constituent trait of borderline personality disorder between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (not all characteristic of my way of being) to 10 (completely characteristic of my way of being) | At 6 months after the intervention
  Evaluation and comparison of the evolution of intensity of each constituent trait of borderline personality disorder between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of suicidal symptomatology (Likert scales from 0 (not all characteristic of my way of being) to 10 (completely characteristic of my way of being) | At 12 months after the intervention
  Evaluation and comparison of the evolution of intensity of each constituent trait of borderline personality disorder between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of para- suicidal symptomatology using the Columbia Suicide Severity Rating Scale (C-SSRS) | At one week after the intervention
  Evaluation and comparison of para -suicidal symptomatology between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 17 close-ended questions of the Columbia-Suicide severity rating scale
Evolution of para- suicidal symptomatology using the Columbia Suicide Severity Rating Scale (C-SSRS) | At 6 months after the intervention
  Evaluation and comparison of para -suicidal symptomatology between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)with the 17 close-ended questions of the Columbia-Suicide severity rating scale
Evolution of para- suicidal symptomatology using the Columbia Suicide Severity Rating Scale (C-SSRS) | At 12 months after the intervention
  Evaluation and comparison of para -suicidal symptomatology between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 17 close-ended questions of the Columbia-Suicide severity rating scale
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At one week after the intervention
  Evaluation and comparison of suicidal symptomatology between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At 6 months after the intervention
  Evaluation and comparison of suicidal symptomatology between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At 12 months after the intervention
  Evaluation and comparison of suicidal symptomatology between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal intensity of suicidal intent) | At one week after the intervention
  Evaluation and comparison of intensity of suicidal intent between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal intensity of suicidal intent) | At 6 months after the intervention
  Evaluation and comparison of intensity of suicidal intent between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal intensity of suicidal intent) | At 12 months after the intervention
  Evaluation and comparison of intensity of suicidal intent between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal intensity of imperious need for non-suicidal self-damaging behavior) | At one week after the intervention
  Evaluation and comparison of intensity of imperious need for non-suicidal self-damaging behavior between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal intensity of imperious need for non-suicidal self-damaging behavior) | At 6 months after the intervention
  Evaluation and comparison of intensity of imperious need for non-suicidal self-damaging behavior between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal intensity of imperious need for non-suicidal self-damaging behavior) | At 12 months after the intervention
  Evaluation and comparison of intensity of imperious need for non-suicidal self-damaging behavior between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal quality of perceived social support) | At one week after the intervention
  Evaluation and comparison of quality of perceived social support between pre-intervention and post-intervention (one week after the last session of the intervention)within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal quality of perceived social support) | At 6 months after the intervention
  Evaluation and comparison of quality of perceived social support between pre-intervention and post-intervention (one week after the last session of the intervention)within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal quality of perceived social support) | At 12 months after the intervention
  Evaluation and comparison of quality of perceived social support between pre-intervention and post-intervention (one week after the last session of the intervention)within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal psychological pain) | At one week after the intervention
  Evaluation and comparison of psychological pain between pre-intervention and post-intervention (one week after of the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal psychological pain) | At 6 months after the intervention
  Evaluation and comparison of psychological pain between pre-intervention and post-intervention (one week after of the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (none) to 10 (maximal psychological pain) | At 12 months after the intervention
  Evaluation and comparison of psychological pain between pre-intervention and post-intervention (one week after of the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (not all characteristic of my way of being) to 10 (completely characteristic of my way of being) | At one week after the intervention
  Evaluation and comparison of the evolution of intensity of each constituent trait of borderline personality disorder between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (not all characteristic of my way of being) to 10 (completely characteristic of my way of being) | At 6 months after the intervention
  Evaluation and comparison of the evolution of intensity of each constituent trait of borderline personality disorder between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of para-suicidal symptomatology (Likert scales from 0 (not all characteristic of my way of being) to 10 (completely characteristic of my way of being) | At 12 months after the intervention
  Evaluation and comparison of the evolution of intensity of each constituent trait of borderline personality disorder between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)
Evolution of the borderline symptomatology using the Borderline Symptom List-23 (BSL-23) scale | At one week after the intervention
  Evaluation and comparison of the evolution of the borderline symptomatology between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 24 items of the Borderline Symptom List-23 (BSL-23) scale. For every question, the subject has to choose a score from 0 to 4 (from not at all to very strongly)
Evolution of the borderline symptomatology using the Borderline Symptom List-23 (BSL-23) scale | At 6 months after the intervention
  Evaluation and comparison of the evolution of the borderline symptomatology between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 24 items of the has to choose a score from 0 to 4 (from not at all to very strongly)
Evolution of the borderline symptomatology using the Borderline Symptom List-23 (BSL-23) scale | At 12 months after the intervention
  Evaluation and comparison of the evolution of the borderline symptomatology between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 24 items of the Borderline Symptom List-23 (BSL-23) scale. For every question, the subject has to choose a score from 0 to 4 (from not at all to very strongly)
Evolution of emotional regulation abilities using the Difficulties in Emotion Regulation Scale (DERS) | At one week after the intervention
  Evaluation and comparison of the evolution of emotional regulation abilities between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 36 items of the Difficulties in Emotion Regulation Scale. For every question, the subject has to choose a score from 1 to 5 (from almost never to almost always)
Evolution of emotional regulation abilities using the Difficulties in Emotion Regulation Scale (DERS) | At 6 months after the intervention
  Evaluation and comparison of the evolution of emotional regulation abilities between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 36 items of the Difficulties in Emotion Regulation Scale. For every question, the subject has to choose a score from 1 to 5 (from almost never to almost always)
Evolution of emotional regulation abilities using the Difficulties in Emotion Regulation Scale (DERS) | At 12 months after the intervention
  Evaluation and comparison of the evolution of emotional regulation abilities between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 36 items of the Difficulties in Emotion Regulation Scale. For every question, the subject has to choose a score from 1 to 5 (from almost never to almost always)
Evolution of propensity to dissociation using the Dissociative Experience Scale (DES) | At one week after the intervention
  Evaluation and comparison of the propensity to dissociation between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 28 items of the Dissociative Experience Scale. For every question, the subject has to choose a score from 0% to 100%.
Evolution of propensity to dissociation using the Dissociative Experience Scale (DES) | At 6 months after the intervention
  Evaluation and comparison of the propensity to dissociation between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 28 items of the Dissociative Experience Scale. For every question, the subject has to choose a score from 0% to 100%.
Evolution of propensity to dissociation using the Dissociative Experience Scale (DES) | At 12 months after the intervention
  Evaluation and comparison of the propensity to dissociation between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 28 items of the Dissociative Experience Scale. For every question, the subject has to choose a score from 0% to 100%.
Anxiety state using the State-Trait Anxiety Inventory (STAI-Trait) | At one week after the intervention
  Evaluation and comparison of the state of anxiety between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 20 items of the State-Trait Anxiety Inventory (STAI-Trait). For every question, the subject has to choose a score from 0 to 3 (from almost never to almost always)
Anxiety state using the State-Trait Anxiety Inventory (STAI-Trait) | At 6 months after the intervention
  Evaluation and comparison of the state of anxiety between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 20 items of has to choose a score from 0 to 3 (from almost never to almost always)
Anxiety state using the State-Trait Anxiety Inventory (STAI-Trait) | At 12 months after the intervention
  Evaluation and comparison of the state of anxiety between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 20 items of the State-Trait Anxiety Inventory (STAI-Trait). For every question, the subject has to choose a score from 0 to 3 (from almost never to almost always)
Anxiety state using the State-Trait Anxiety Inventory (STAI-State) | At one week after the intervention
  Evaluation and comparison of the state of anxiety between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT)with the 20 items of the State-Trait Anxiety Inventory (STAI-State). For every question, the subject has to choose a score from 0 to 3 (from no to yes)
Anxiety state using the State-Trait Anxiety Inventory (STAI-State) | At 6 months after the intervention
  Evaluation and comparison of the state of anxiety between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 20 items of the State-Trait Anxiety Inventory (STAI-State). For every question, the subject has to choose a score from 0 to 3 (from no to yes)
Anxiety state using the State-Trait Anxiety Inventory (STAI-State) | At 12 months after the intervention
  Evaluation and comparison of the state of anxiety between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (DBT versus DBT+ACT) with the 20 items of the State-Trait Anxiety Inventory (STAI-State). For every question, the subject has to choose a score from 0 to 3 (from no to yes)
Anger state using the Spielberger State-Trait Anger Expression Inventory (STAXI-TRAIT) | At 6 months after the intervention
  Evaluation and comparison of the state of anger between pre-intervention and 6 months post-intervention within the two groups (DBT versus DBT+ACT) with the 33 items of Spielberger State-Trait Anger Expression Inventory (STAXI-TRAIT). For every question, the subject has to choose a score from 1 to 4 (from almost never to almost always)
Anger state using the Spielberger State-Trait Anger Expression Inventory (STAXI-TRAIT) | At 12 months after the intervention
  Evaluation and comparison of the state of anger between pre-intervention and 6 months post-intervention within the two groups (DBT versus DBT+ACT) with the 33 items of Spielberger State-Trait Anger Expression Inventory (STAXI-TRAIT). For every question, the subject has to choose a score from 1 to 4 (from almost never to almost always)
Anger state using the Spielberger State-Trait Anger Expression Inventory (STAXI-ETAT) | At one week after the intervention
  Evaluation and comparison of the state of anger between pre-intervention and 6 months post-intervention within the two groups (DBT versus DBT+ACT) with the 10 items of Spielberger State-Trait Anger Expression Inventory (STAXI-ETAT). For every question, the subject has to choose a score from 1 to 4 (from not at all to a lot)
Anger state using the Spielberger State-Trait Anger Expression Inventory (STAXI-ETAT) | At 6 months after the intervention
  Evaluation and comparison of the state of anger between pre-intervention and 6 months post-intervention within the two groups (DBT versus DBT+ACT) with the 10 items of Spielberger State-Trait Anger Expression Inventory (STAXI-ETAT). For every question, the subject has to choose a score from 1 to 4 (from not at all to a lot)
Anger state using the Spielberger State-Trait Anger Expression Inventory (STAXI-ETAT) | At 12 months after the intervention
  Evaluation and comparison of the state of anger between pre-intervention and 6 months post-intervention within the two groups (DBT versus DBT+ACT) with the 10 items of Spielberger State-Trait Anger Expression Inventory (STAXI-ETAT). For every question, the subject has to choose a score from 1 to 4 (from not at all to a lot)
Hopelessness using the Beck Hopelessness Scale (BHS) | At one week after the intervention
  Evaluation and comparison of the hopelessness between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 20 items of the Beck Hopelessness Scale. For every question, the subject has to answer true or false
Hopelessness using the Beck Hopelessness Scale (BHS) | At 6 months after the intervention
  Evaluation and comparison of the hopelessness between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 20 items of the Beck Hopelessness Scale. For every question, the subject has to answer true or false
Hopelessness using the Beck Hopelessness Scale (BHS) | At 12 months after the intervention
  Evaluation and comparison of the hopelessness between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 20 items of the Beck Hopelessness Scale. For every question, the subject has to answer true or false.
Quality Of Life evaluated by the World Health Organization Quality of Life measure (WHOQOL-BREF) | At one week after the intervention
  Evaluation and comparison of the quality of life between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 20 items of the World Health Organization Quality of Life measure (WHOQOL-BREF). For every question, the subject has to choose a score from 1 to 5.
Quality Of Life evaluated by the World Health Organization Quality of Life measure (WHOQOL-BREF) | At 6 months after the intervention
  Evaluation and comparison of the quality of life between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 20 items of the World Health Organization Quality of Life measure (WHOQOL-BREF). For every question, the subject has to choose a score from 1 to 5.
Quality Of Life evaluated by the World Health Organization Quality of Life measure (WHOQOL-BREF) | At 12 months after the intervention
  Evaluation and comparison of the quality of life between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 20 items of the World Health Organization Quality of Life measure (WHOQOL-BREF). For every question, the subject has to choose a score from 1 to 5.
Acceptance assessment using the Acceptance and Action Questionnaire (AAQII) | At one week after the intervention
  Evaluation and comparison of the acceptance between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 10 items of the Acceptance and Action Questionnaire (AAQII)). For every question, the subject has to choose a score from 1 to 7(never true to always true).
Acceptance assessment using the Acceptance and Action Questionnaire (AAQII) | At 6 months after the intervention
  Evaluation and comparison of the acceptance between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 10 items of the Acceptance and Action Questionnaire (AAQII)). For every question, the subject has to choose a score from 1 to 7(never true to always true).
Acceptance assessment using the Acceptance and Action Questionnaire (AAQII) | At 12 months after the intervention
  Evaluation and comparison of the acceptance between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 10 items of the Acceptance and Action Questionnaire (AAQII)). For every question, the subject has to choose a score from 1 to 7(never true to always true).
Contact with the present moment assessment using the Mindful Attention Awareness Scale (MAAS) | At one week after the intervention
  Evaluation and comparison of the contact with the present moment between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 15 items of Mindful Attention Awareness Scale (MAAS). For every question, the subject has to choose a score from 1 to 6 (almost always to almost never).
Contact with the present moment assessment using the Mindful Attention Awareness Scale (MAAS) | At 6 months after the intervention
  Evaluation and comparison of the contact with the present moment between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 15 items of Mindful Attention Awareness Scale (MAAS). For every question, the subject has to choose a score from 1 to 6 (almost always to almost never).
Contact with the present moment assessment using the Mindful Attention Awareness Scale (MAAS) | At 12 months after the intervention
  Evaluation and comparison of the contact with the present moment between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 15 items of Mindful Attention Awareness Scale (MAAS). For every question, the subject has to choose a score from 1 to 6 (almost always to almost never).
Meaning in life assessment using Life Regard Index (LRI) | At one week after the intervention
  Evaluation and comparison of the contact with the present moment between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 28 items of the Life Regard Index (LRI)). For every question, the subject has to answer agree, neutral or ont agree
Meaning in life assessment using Life Regard Index (LRI) | At 6 months after the intervention
  Evaluation and comparison of the contact with the present moment between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 28 items of the Life Regard Index (LRI)). For every question, the subject has to answer agree, neutral or ont agree
Meaning in life assessment using Life Regard Index (LRI) | At 12 months after the intervention
  Evaluation and comparison of the contact with the present moment between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the 28 items of the Life Regard Index (LRI)). For every question, the subject has to answer agree, neutral or ont agree
Satisfaction of the intervention using the Likert scales rating from 0 (not at all satisfied) to 10 (extremely satisfied) | At one week after the intervention
  Evaluation of the satisfaction about the intervention within the two groups (DBT versus DBT+ACT)
Quality of life related to health using the EQ5D-3L questionnaire | At 6 months after the intervention
  Evaluation and comparison of the quality of life between pre-intervention and 6 months post-intervention within the two groups (DBT versus DBT+ACT) with the 5 items of the EQ5D-3L. For every question, the subject has the choice between 3 answers.
Quality of life related to health using the EQ5D-3L questionnaire | At 12 months after the intervention
  Evaluation and comparison of the quality of life between pre-intervention and 6 months post-intervention within the two groups (DBT versus DBT+ACT) with the 5 items of the EQ5D-3L. For every question, the subject has the choice between 3 answers.
Depression intensity using the Inventory of Depressive Symptomatology (IDS-C30) | At one week after the intervention
  Evaluation and comparison of the intensity of depression between pre-intervention and post-intervention (one week after the last session) within the two groups (DBT versus DBT+ACT) with the 30 items of Inventory of Depressive Symptomatology (IDS-C30). For every item corresponding to a depressive symptom, the investigator has the choice between 3 levels of response.
Depression intensity using the Inventory of Depressive Symptomatology (IDS-C30) | At 6 months after the intervention
  Evaluation and comparison of the intensity of depression between pre-intervention and post-intervention (one week after the last session) within the two groups (DBT versus DBT+ACT) with the 30 items of Inventory of Depressive Symptomatology (IDS-C30). For every item corresponding to a depressive symptom, the investigator has the choice between 3 levels of response.
Depression intensity using the Inventory of Depressive Symptomatology (IDS-C30) | At 12 months after the intervention
  Evaluation and comparison of the intensity of depression between pre-intervention and post-intervention (one week after the last session) within the two groups (DBT versus DBT+ACT) with the 30 items of Inventory of Depressive Symptomatology (IDS-C30). For every item corresponding to a depressive symptom, the investigator has the choice between 3 levels of response.
Global functioning using the Global Assessment of Functioning Scale (GAF) | At one week after the intervention
  Evaluation and comparison of the global functioning between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the Global Assessment of Functioning Scale (GAF).With this scale, the investigator has to give a score between 0 to 100 for the global functioning of the patient
Global functioning using the Global Assessment of Functioning Scale (GAF) | At 6 months after the intervention
  Evaluation and comparison of the global functioning between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the Global Assessment of Functioning Scale (GAF).With this scale, the investigator has to give a score between 0 to 100 for the global functioning of the patient
Global functioning using the Global Assessment of Functioning Scale (GAF) | At 12 months after the intervention
  Evaluation and comparison of the global functioning between pre-intervention and post-intervention (one week after the intervention) within the two groups (DBT versus DBT+ACT) with the Global Assessment of Functioning Scale (GAF).With this scale, the investigator has to give a score between 0 to 100 for the global functioning of the patient
Incremental cost-effectiveness ratio (ICER) | At 1 year follow-up
  Evaluation and comparison of the incremental cost-effectiveness ratio between pre-intervention and 12 months post-intervention within the two groups (DBT versus DBT+ACT)
Incremental cost-utility ratio (ICUR) | At 1 year follow-up
  Evaluation and comparison of the incremental cost-utility ratio between pre-intervention and 12 months post-intervention within the two groups (DBT versus DBT+ACT)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, Hérault, France